CLINICAL TRIAL: NCT03289104
Title: Improving Sternal Healing After Cardiac Surgery: Sternal Wire vs ZIPFIX
Acronym: Closure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to inadequate funding.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Marc Ruel MD MPH FRCSC, Chief Cardiac Surgeon, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160921
Record Dates: First submitted 2017-01-31; First posted 2017-09-20 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Sternal Injury; Cardiac Surgery; Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steel Wires (Active Comparator): In this arm, patients will have their sternum closed with steel wires.
  Interventions: Device: Steel Wires
- ZipFix Sternal Closure System (Plastic Cables) (Experimental): In this arm, patients will have their sternum closed with the ZipFix system.
  Interventions: Device: ZipFix Sternal Closure System

INTERVENTIONS:
Device: Steel Wires — Control: Steel wires (device) are selected for sternal closure after surgery. Currently, most patients who have a sternotomy during cardiac surgery have their sternum closed with steel wires.
  Arms: Steel Wires
Device: ZipFix Sternal Closure System — Treatment: ZipFix system (device) are selected for sternal closure after surgery. These plastic cables can also be used to close the sternum during bypass surgery.
  Arms: ZipFix Sternal Closure System (Plastic Cables)

SUMMARY:
The objective of this study is to determine whether sternal reconstruction using the ZIPFIX system compared to standard wire cerclage could improve bone healing, patient function, and decreased postoperative pain.

DETAILED DESCRIPTION:
Despite a longer time for bone healing and functional recovery, median sternotomy is still the most common approach in cardiac surgery. Sternal closure has traditionally been wire cerclage using stainless steel wires, however, new sternal fixation devices have been developed to improve sternal union. Rigid sternal fixation, although very costly, has demonstrated to be superior to standard wire cerclage both in clinical and biomechanical studies. Although improved sternal healing was observed with rigid plate fixation in a randomized controlled trial in high risk patients, the wound complication rate with plate fixation was almost double that of wire cerclage albeit not statistically significant.

A novel sternal closure system denoted the sternal ZIPFIX system (DePuySynthes, Companies of Johnson and Johnson, West Over, PA, US) is biocompatible Poly-Ether-Ether-Ketone implant that was developed for fast and reliable sternal fixation following median sternotomy. First published case series utilized the sternal ZIPFIX System demonstrating effective sternal stability at 30 days. Another study has demonstrated no significant difference in the incidence of sternal wound infection following the ZIPFIX system compared to standard wire cerclage while Stelly et al., 2015 demonstrated reduced risk of deep sternal wound infection for patients using ZIPFIX. The ZIPFIX system demonstrates a higher resistance of fatigue failure and has a larger implant-to-bone contact area compared to stainless steel wires thereby reducing the risk of bone cut through. Placement of the cable ties are done similar to wire cerclage thereby not affecting time for sternal closure and training.

The objective of this study is to determine whether sternal reconstruction using the ZIPFIX system compared to standard wire cerclage would improve bone healing, patient function, and decrease postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Scheduled cardiac surgery including coronary artery bypass grafting, aortic valve replacement, mitral valve replacement/repair, or ascending aorta replacement.
* Patient undergoing elective or urgent surgery
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Patients undergoing emergent cardiac surgery
* Severe congestive heart failure (NYHA class III or IV) at enrollment
* Prior cardiac surgery
* Patients undergoing ventricular assist device insertion or heart transplantation
* Patients with a known metal allergy or allergy to ZIPFIX implant
* Patients who refuses consent
* Patients who are unable to follow post-operative instructions
* Prior history of significant bleeding that might be expected to recur with cardiac surgery
* Dementia with a mini mental status examination (MMSE) score of < 20
* Extra cardiac illness that is expected to limit survival to less than 5 years
* Suspected pregnancy. A pregnancy test (urine or serum) will be administered to all women not clearly menopausal
* Concurrent enrollment in another clinical trial
* Geographic inaccessibility for follow-up visits required by the protocol
* Prisoners or institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Sternal bone healing | 3 months after surgery
  Assessment of how the sternum is healing, assessed via a CT scan and classified using a 6-point scale.

SECONDARY OUTCOMES:
Post-operative pain | Within 1 week of surgery
  A patient's subjective assessment of their pain after surgery.
Use of narcotics | In the first 6 months after surgery
  A patient's use of narcotic pain medication. To assess this measure, the proportion of patients in each group using narcotic pain medication will be compared.
Sternal instability | In the first 6 months after surgery
  Clinical assessment of patient's sternum stability after surgery
Sternal wound infection | In the first 6 months after surgery
  The presence of sternal wound infection after surgery, confirmed by wound cultures
Cost | In the first 6 months after surgery.
  An approximation of the comparative cost of the ZipFix system versus sternal wires, which will be approximated by comparing the duration of hospital stay between groups; the use of narcotic pain medication between groups; and the rate of sternal wound infection between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD, MPH, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- Division of Cardiac Surgery, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karamlou T, Jacobs ML, Pasquali S, He X, Hill K, O'Brien S, McMullan DM, Jacobs JP. Surgeon and center volume influence on outcomes after arterial switch operation: analysis of the STS Congenital Heart Surgery Database. Ann Thorac Surg. 2014 Sep;98(3):904-11. doi: 10.1016/j.athoracsur.2014.04.093. Epub 2014 Jul 25. PMID 25069686
- [Background] Kozower BD, Sheng S, O'Brien SM, Liptay MJ, Lau CL, Jones DR, Shahian DM, Wright CD. STS database risk models: predictors of mortality and major morbidity for lung cancer resection. Ann Thorac Surg. 2010 Sep;90(3):875-81; discussion 881-3. doi: 10.1016/j.athoracsur.2010.03.115. PMID 20732512
- [Background] Raman J, Song DH, Bolotin G, Jeevanandam V. Sternal closure with titanium plate fixation--a paradigm shift in preventing mediastinitis. Interact Cardiovasc Thorac Surg. 2006 Aug;5(4):336-9. doi: 10.1510/icvts.2005.121863. Epub 2006 Apr 25. PMID 17670585
- [Background] Pai S, Gunja NJ, Dupak EL, McMahon NL, Roth TP, Lalikos JF, Dunn RM, Francalancia N, Pins GD, Billiar KL. In vitro comparison of wire and plate fixation for midline sternotomies. Ann Thorac Surg. 2005 Sep;80(3):962-8. doi: 10.1016/j.athoracsur.2005.03.089. PMID 16122464
- [Background] Losanoff JE, Basson MD, Gruber SA, Huff H, Hsieh FH. Single wire versus double wire loops for median sternotomy closure: experimental biomechanical study using a human cadaveric model. Ann Thorac Surg. 2007 Oct;84(4):1288-93. doi: 10.1016/j.athoracsur.2007.05.023. PMID 17888985
- [Background] Losanoff JE, Collier AD, Wagner-Mann CC, Richman BW, Huff H, Hsieh Fh, Diaz-Arias A, Jones JW. Biomechanical comparison of median sternotomy closures. Ann Thorac Surg. 2004 Jan;77(1):203-9. doi: 10.1016/s0003-4975(03)01468-1. PMID 14726062
- [Background] Song DH, Lohman RF, Renucci JD, Jeevanandam V, Raman J. Primary sternal plating in high-risk patients prevents mediastinitis. Eur J Cardiothorac Surg. 2004 Aug;26(2):367-72. doi: 10.1016/j.ejcts.2004.04.038. PMID 15296898
- [Background] Grapow MT, Melly LF, Eckstein FS, Reuthebuch OT. A new cable-tie based sternal closure system: description of the device, technique of implantation and first clinical evaluation. J Cardiothorac Surg. 2012 Jun 25;7:59. doi: 10.1186/1749-8090-7-59. PMID 22731778
- [Background] Melly L, Gahl B, Meinke R, Rueter F, Matt P, Reuthebuch O, Eckstein FS, Grapow MT. A new cable-tie-based sternal closure device: infectious considerations. Interact Cardiovasc Thorac Surg. 2013 Aug;17(2):219-23; discussion 223-4. doi: 10.1093/icvts/ivt183. Epub 2013 Apr 26. PMID 23624983
- [Background] Stelly MM, Rodning CB, Stelly TC. Reduction in deep sternal wound infection with use of a peristernal cable-tie closure system: a retrospective case series. J Cardiothorac Surg. 2015 Nov 14;10:166. doi: 10.1186/s13019-015-0378-7. PMID 26577944